CLINICAL TRIAL: NCT02680028
Title: Randomised Trial of Trochanteric Hip Fractures Treated With Either a Short or Standard Length Intramedullary Nail
Brief Title: Short Versus Standard Intramedullary Nail for Trochanteric Hip Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peterborough and Stamford Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Martyn J Parker, Consultant Orthopaedic Surgeon, Peterborough and Stamford Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R&D/2015/28
Record Dates: First submitted 2016-02-04; First posted 2016-02-11 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard length intramedullary nail (Active Comparator): 220mm intramedullary nail
  Interventions: Device: targon pft nail
- Short length intramedullary nail (Experimental): 175mm intramedullary nail
  Interventions: Device: targon pft nail

INTERVENTIONS:
Device: targon pft nail — 220 mm vs 175mm nail

SUMMARY:
In England each year over 65,000 people fracture their hip. Most of these patients are elderly females with the fracture occurring after a simple trip or stumble. Approximately half of these fractures are classified from their relationship to the hip joint capsule as extracapsular. The majority of these fractures are treated surgically by internal fixation using, either a plate and screws (sliding hip screw) or nail and screws (intramedullary nail).

Recent randomised studies from Peterborough involving 1000 patients have indicated that there are modest benefits for treating this type of fracture with an intramedullary nail in comparison to a sliding hip screw. This study aims to progress from these earlier studies to determine if a slightly thinner and shorter intramedullary nail (175mm in length), has any significant advantages or disadvantages to the standard length (220mm) intramedullary nail.

Both implants to be used in this study are in routine use around the world and are being used within their licenced indication. The study is therefore using two different designs of implant within their recommended area of use, but in which there is uncertainty as to which is the best design.

DETAILED DESCRIPTION:
The trial will be run as close to the ideal trial methodology for a randomised trial as specified by the CONSORT statement as possible. This will include secure randomisation, intention to treat analysis, full reporting of outcomes and clinical follow-up by a person who is blinded to the prosthesis used. The trial will follow the code of good clinical practice as specified by the hospital trusts Research and Development Committee.

In Peterborough all hip fracture patients are admitted to the acute trauma ward and transferred to the care of the Chief Investigator (Mr Martyn Parker (MJP)). Those patients that are willing to participant in this randomised trial are consented prior to surgery. Treatment follows standard evidence based protocols with follow-up of all patients in a hip fracture clinic. A comprehensive database is maintained for all patients containing both audit and research data. Included in this is a standardised assessment of outcome.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to Peterborough City Hospital with a trochanteric hip fracture (type A1 type A2) that is to be treated by internal fixation with an intramedullary nail.

Exclusion Criteria:

* Patients who decline to participate or in whom consent or assent is not available

  * Patients admitted when MJP is not available to supervise treatment
  * Patients with pathological fractures from Paget's disease of bone secondaries from tumour
  * Patients with a Subtrochanteric fracture and those of the reversed and transverse fracture type (A3 fractures)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Regain of mobility as assessed by a mobility score | 1 year
  Parker MJ, Palmer CR. A new mobility score for predicting mortality after hip fracture. J Bone Joint Surg Br. 1993;75:797-8.
  Validation Kristensen MT, Bandholm T, Foss NB, Ekdahl C, Kehlet H. High inter-tester reliability of the new mobility score in patients with hip fracture. J Rehabil Med 2008;40:589-91.
  Mobility will be assessed using a scale of 0 to 9. Nine represents full mobility indoors and outdoors without walking aids; Zero represents a bed-bound patient.

CONTACTS AND LOCATIONS:
Overall Officials: martyn parker, Principal Investigator — Peterborough hospital nhs trust
Locations (1):
- Peterbrough City Hospital, Peterborough, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Parker MJ, Cawley S. Short (175 mm) versus standard (220 mm) length intramedullary nail for trochanteric hip fractures: a randomized trial of 229 patients. Bone Joint J. 2020 Mar;102-B(3):394-399. doi: 10.1302/0301-620X.102B3.BJJ-2019-0776.R3. PMID 32114812